CLINICAL TRIAL: NCT06139822
Title: Effects of Hamstring Stretching With Conventional Physical Therapy in Plantar Fasciitis
Brief Title: Hamstring Stretching in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/RCRS/01223 Sunya Fiaz
Record Dates: First submitted 2023-01-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Plantar Fasciitis of Both Feet
Keywords: Planter Faciatis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): hamstring stretching, cold pack, stretching, strengthening of plantar fascia and calf muscles.
  . Hamstring stretching will be used as an intervention protocol along with conventional physical therapy. Treatment protocol will be followed for thrice a week for 2 weeks. The session will be of approximately 20 minutes. Patient will be in supine lying, passively increase hip flexion while keeping the back straight, and the knee in the extended position from the start to the end of the stretching while the ankle will be in a neutral position
  a 30-second rest period will be recommended between stretching repetitions. For each stretching repetition, the individual had to achieve a position of mild discomfort (not pain) which will sustain for 30 seconds.
  Interventions: Other: Experimental Group
- Control Group (Active Comparator): Cold pack, stretching, strengthening of plantar fascia and calf muscles
  Control group included Cold pack for 7 to 10 mins. Followed by stretching of plantar fascia through:
  * toe stretches to stretch the plantar fascia.
  * towel to stretch the bottom of foot (towel scrunches)
  * calf muscles stretching
  After stretching exercises strengthening is performed by the following:
  * towel curls
  * heel raise Patients performed 2 sets, each repetition lasting 30 seconds, 2 times a day for each exercise.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Hamstring stretching is the main intervention which is being used along with convention protocol for plantar fasciitis.
  Other Names: Hamstring Streching
  Arms: Experimental Group
Other: Control Group — Control group included Cold pack for 7 to 10 mins. Followed by stretching of plantar fascia .
  Other Names: cold pack, calf and plantar fascia stretchings and strenthening exercises
  Arms: Control Group

SUMMARY:
The purpose of the study is to compare the effects of Hamstring stretching versus conventional treatment for plantar fasciitis. A randomized control trial was conducted at Cena Medical Center Rawalpindi and Midland Doctors Institute Muzaffarabaad. The sample size was 64 calculated through open-epi tool. The participants were divided into two groups, interventional and control group each having 32 participants. The study duration was 1 year. Sampling technique applied was Purposive sampling for recruitment and group randomization using flip coin method. Only 25to 45 years participants with plantar fasciitis along with hamstring tightness were included in the study. Tools used in this study are Goniometer, Visual Analogue Scale(VAS) for pain, and Functional Foot Index (FFI) for pain and disability. Data was collected before treatment at baseline and after 1st and 2nd week of the application of interventions. Data analyzed through SPSS version 25.

DETAILED DESCRIPTION:
Plantar fasciitis is one of the main causes of heel pain. it is caused by the micro trauma to the site of attachment of plantar fascia at its origin on the medial tubercle of calcaneus resulting in inflammation. Plantar fascia is a fibrous band present at the bottom of foot which attaches heel to each of the toes.plantar fascia has a windlass mechanism which continuously stretches and shortens facilitating foot movements during walk.

During the standing phase all the tension forces are gathered at calcaneal tuberosity, which is a site of attachment for plantar fascia on heel. Pain is generally present at the medial side of heel to the medial arch of the foot.

Plantar fasciitis is often caused in people who have long periods of standing, involved in activities like running, jumping or other repeated activities. After knowing the exact mechanism it is suggested that it should be termed as planter fasciosis.Plantar fasciitis accounts for almost 80% of the total heel pain experienced by the people.

Planter fasciitis is treated with various treatment options. Initially it is treated by conservative treatments such as, rest, ice massage, foot ware modification, oral analgesics, stretching techniques, physical therapy modalities, and night splinting. If pain do not resolve with conservative treatment then further treatment options will be extracorporeal shock wave therapy, cortisone injections and surgery.

Diana et al concluded that addition of manual techniques for trigger point release along with stretching of plantar fascia is more effective than stretching alone. In a randomized control trial with a follow up of 12 months high load strength training was found to be quicker and more efficient treatment for plantar fasciitis. another RCT conducted in 2017 reported that stretching of Achilles tendon along with plantar fascia is twice effective than only plantar fascia stretching.

Immobilization done by using splints at night is one of the best treatments to avoid contracture in plantar fascia during night. But they are also related to sleep disturbances and discomfort during night. By using night splint there has been a pain relief for shorter period of time. Night splints used alongside custom foot orthotics have better results than used alone. Controlled Ankle Movement is very effective in reducing pain in heel. It can be done by using walking boots and casts. These boots and casts will help to reduce over stretching of plantar fascia with unloading mechanism over heel. The reported reduction of pain by this mechanism of controlled ankle movement is in up to 40% of individuals.

Jonathan et al reported that there is a role of hamstring tightness in plantar fasciitis. A correlation study found a strong relationship between hamstring tightness and plantar fasciitis. patients having hamstring tightness are 8.7% more prone towards developing planter fasciitis.

Hamstring is found to be affected in patients with plantar fasciitis. Many studies found relationship of hamstring tightness with plantar fasciitis. Hamstring tightness affects the posterior muscles increasing load on plantar fascia. There is scarce evidence about the hamstring stretching in patients having plantar fasciitis. So this study will focus on hamstring stretching along with plantar fascia stretching and strengthening to improve pain, range of motion and disability.

ELIGIBILITY:
Inclusion Criteria:

1. Both Genders
2. 25 to 45 years of age
3. Participants having heel pain for more than one month.
4. Participants having Windlass positive test.
5. Participants having hamstring tightness.
6. sit and reach test positive.
7. Bilateral plantar fasciitis.

Exclusion Criteria:

* Patients with corticosteroid injection
* Fracture around ankle and Calcaneal
* Any soft tissue injuries around ankle.
* Other Neurological/ Musculoskeletal disorder
* Congenital foot anomalies
* Systemic medical illness

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | upto 2 weeks
  The visual analogue scale (VAS) is a scale that is used as a questionnaire. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end points.patient rates its pain between 0 to 10.
  VAS Visual Analogue Scale changes measured at baseline after 1 week and sfter 2nd week.

SECONDARY OUTCOMES:
Goniometery for ROM(Range of Motion) | upto 2 weeks
  The art and science of measuring the joint ranges in each plane of the joint are called goniometry. Goiniometer is used to measure ankle range of motions specifically dorsiflexion and plantar flexion.
  Changes from the Baseline ROM range of Motion of ankle in plantar flexion was taken with the Help of goniometer. Changes from the Baseline ROM range of Motion of ankle in plantar flexion was taken with the Help of goniometer and after 1st and 2nd week
Functional Foot Index (FFI-R) | upto 2 weeks
  A Foot Function Index (FFI-R) was developed to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI-R is a self-administered index consisting of 68 items divided into 4 sub-scales. Both total and sub-scale scores are produced.
  Functional Foot Index (FFI-R) is used to measure activity status and disability index at baseline and after every week.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No